CLINICAL TRIAL: NCT02601573
Title: A Phase II, Randomized, Open-Label Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of Elbasvir/Grazoprevir (EBR/GZR) and Sofosbuvir (SOF) With and Without Ribavirin (RBV) in Cirrhotic Subjects With Chronic HCV GT3 Infection
Brief Title: Elbasvir/Grazoprevir (EBR/GZR) and Sofosbuvir (SOF) With and Without Ribavirin (RBV) in Cirrhotic Subjects With Chronic Hepatitis C Virus (HCV) Genotype 3 (GT3) Infection (MK-5172-083)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-083; 2015-003187-37 (EudraCT Number); MK-5172-083 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir; Ribavirin; Sofosbuvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks (Experimental): TN HCV GT3 participants will take 1 fixed-dose combination (FDC) tablet containing EBR 50 mg+GZR 100 mg and 1 tablet containing SOF 400 mg once-daily (q.d.) with RBV (200 mg capsules; weight-based dosing) twice-daily (b.i.d.) for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin; Drug: Sofosbuvir
- Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks (Experimental): TN HCV GT3 participants will take 1 FDC tablet containing EBR 50 mg+GZR 100 mg and 1 tablet containing SOF 400 mg q.d. for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Sofosbuvir
- Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks (Experimental): TE HCV GT3 participants will take 1 FDC tablet containing EBR 50 mg+GZR 100 mg and 1 tablet containing SOF 400 mg q.d. for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Sofosbuvir
- Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks (Experimental): TE HCV GT3 participants will take 1 FDC tablet containing EBR 50 mg+GZR 100 mg and 1 tablet containing SOF 400 mg q.d. with RBV (200 mg capsules; weight-based dosing) b.i.d. for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Ribavirin; Drug: Sofosbuvir
- Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks (Experimental): TE HCV GT3 participants will take 1 FDC tablet containing EBR 50 mg+GZR 100 mg and 1 tablet containing SOF 400 mg q.d. for 16 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Grazoprevir — GZR 100 mg is a component of the MK-5172A FDC tablet (also containing EBR 50 mg) and was taken q.d. by mouth in the morning.
  Other Names: MK-5172
Drug: Elbasvir — EBR 50 mg is a component of the MK-5172A FDC tablet (also containing GZR 100 mg) and was taken q.d. by mouth in the morning.
  Other Names: MK-8742
Drug: Ribavirin — RBV 200 mg capsules taken b.i.d. (morning and evening) by mouth at a total daily dose ranging from 800 mg to 1400 mg (total daily dose was based on participant body weight).
  Other Names: Rebetol®
  Arms: Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks; Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks
Drug: Sofosbuvir — SOF 400 mg tablet taken q.d. by mouth in the morning with food.
  Other Names: Sovaldi®, Harvoni®

SUMMARY:
This is a randomized, multi-site, open-label trial of the co-administration of a fixed-dose combination (FDC) of EBR 50 mg + GZR (100 mg) (EBR/GZR) and SOF 400 mg, with and without RBV, in treatment-naïve (TN) and treatment-experienced (TE) participants with chronic HCV GT3 infection with compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* has HCV RNA (>= 10,000 IU/mL in peripheral blood) at screening
* has documented HCV GT3 (with no evidence of non-typeable or mixed GT infection)
* has compensated cirrhosis of the liver
* has liver imaging within 6 months of Day 1 with no evidence of hepatocellular carcinoma (HCC)
* is either HCV TN or TE (i.e., has documented prior virologic failure or intolerance to peg-interferon/ribavirin)
* is otherwise healthy as determined by medical history, physical examination, electrocardiogram (ECG), and clinical laboratory measurements
* has compensated cirrhosis of the liver
* is TN or TE (i.e., documented prior virologic failure or intolerance to peg-interferon/ribavirin)
* is not of reproductive potential, or agrees to not impregnate a partner or become pregnant for at least 2 weeks prior to the first dose of study drug, and for 7 months after the final dose of study drug (or longer if dictated by local regulations)

Exclusion Criteria:

* has previously received one or more doses of a direct-acting antiviral (DAA)
* has evidence of decompensated liver disease
* is coinfected with hepatitis B (hepatitis B surface antigen [HBsAg] positive)
* has a recent (within 5 years) history of malignancy or is under evaluation for HCC or other suspected malignancy
* is currently or has participated (within past 30 days) in a study with an investigational compound
* has clinically-relevant drug or alcohol abuse within the past 12 months of screening
* is a female and is pregnant or breast-feeding
* is a male whose female partner is/are pregnant
* has any of the following:
* organ transplants
* poor venous access
* history of gastric surgery or malabsorption disorder
* current or history of clinically significant cardiac abnormalities or dysfunction
* chronic pulmonary disease
* hemoglobinopathy
* history of hospitalization within 3 months prior to enrollment
* medical or surgical condition that may result in need for hospitalization during the course of the study
* any condition requiring, or likely to require, chronic systemic administration of corticosteroids, tumor necrosis factor (TNF) antagonists, or other immunosuppresant drugs during the course of the study
* any condition, prestudy laboratory or ECG abnormality, or history of any illness, which could confound results of the study or pose additional risks in administering study drugs in the opinion of the investigator
* has a life-threatening serious AE (SAE) during the screening period
* has evidence of history of chronic hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Foster GR, Agarwal K, Cramp ME, Moreea S, Barclay S, Collier J, Brown AS, Ryder SD, Ustianowski A, Forton DM, Fox R, Gordon F, Rosenberg WM, Mutimer DJ, Du J, Gilbert CL, Asante-Appiah E, Wahl J, Robertson MN, Barr E, Haber B. Elbasvir/grazoprevir and sofosbuvir for hepatitis C virus genotype 3 infection with compensated cirrhosis: A randomized trial. Hepatology. 2018 Jun;67(6):2113-2126. doi: 10.1002/hep.29852. Epub 2018 Apr 19. PMID 29473975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants infected with HCV GT3 were enrolled at 14 study centers in the United Kingdom.
Pre-assignment Details: A total of 101 participants were randomized, including 1 participant who did not meet inclusion criteria and who should have been considered a screen failure; this participant was not treated with study drug. A total of 100 participants were treated.
Groups:
- Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks: Treatment-naïve (TN) Hepatitis C virus (HCV) genotype 3 (GT3) participants took 1 fixed-dose combination (FDC) tablet containing elbasvir (EBR) 50 mg + grazoprevir (GZR) 100 mg and 1 tablet containing sofosbuvir (SOF) 400 mg once daily (q.d.) with ribavirin (RBV) (200 mg capsules; weight-based dosing) twice daily (b.i.d.) for 8 weeks.
- Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks: TN HCV GT3 participants took 1 FDC tablet containing EBR 50 mg + GZR 100 mg and 1 tablet containing SOF 400 mg q.d. for 12 weeks.
- Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks: Treatment-experienced (TE) HCV GT3 participants took 1 FDC tablet containing EBR 50 mg + GZR 100 mg and 1 tablet containing SOF 400 mg q.d. for 12 weeks.
- Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks: TE HCV GT3 participants took 1 FDC tablet containing EBR 50 mg + GZR 100 mg and 1 tablet containing SOF 400 mg q.d. with RBV (200 mg capsules; weight-based dosing) b.i.d. for 12 weeks.
- Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks: TE HCV GT3 participants took 1 FDC tablet containing EBR 50 mg+GZR 100 mg and 1 tablet containing SOF 400 mg q.d. for 16 weeks.
Period: Overall Study
Arm/Group | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks
Started | 23 (Number randomized and treated.) | 24 (Number randomized and treated.) | 17 (Number randomized and treated.) | 18 (Number randomized and treated.) | 18 (Number randomized and treated.)
Completed | 23 | 20 | 16 | 17 | 16
Not Completed | 0 | 4 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 3 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis population includes only the 100 participants who were both randomized and treated.
Groups:
- Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks: TN HCV GT3 participants took 1 FDC tablet containing EBR 50 mg + GZR 100 mg and 1 tablet containing SOF 400 mg q.d. with RBV (200 mg capsules; weight-based dosing) b.i.d. for 8 weeks.
- Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks: TE HCV GT3 participants took 1 FDC tablet containing EBR 50 mg + GZR 100 mg and 1 tablet containing SOF 400 mg q.d. for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks | Total
Number analyzed (Participants) | 23 | 24 | 17 | 18 | 18 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (9.0) | 48.1 (9.3) | 58.6 (6.1) | 56.1 (8.4) | 53.8 (6.4) | 53.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 6 | 6 | 3 | 32
  Male | 13 | 17 | 11 | 12 | 15 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving SVR12 (Sustained Virologic Response 12 Weeks After the End of All Study Therapy)
Description: The percentage of participants achieving SVR12 (i.e., HCV ribnonucleic acid [RNA] < Lower Limit of Quantification [LLOQ] 12 weeks after completing study treatment) was determined. Plasma HCV RNA levels were determined with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay, which has a LLOQ of 15 IU/mL.
Time Frame: Up to Week 28
Population: All randomized participants who received at least 1 dose of study drug, were not lost to follow-up for reasons unrelated to study treatment, and had SVR12 data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks
Number analyzed (Participants) | 23 | 23 | 17 | 17 | 18
Percentage of Participants | 91.3 [72.0 to 98.9] | 100.0 [85.2 to 100.0] | 100.0 [80.5 to 100.0] | 100.0 [80.5 to 100.0] | 94.4 [72.7 to 99.9]

2. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 18 weeks (up to 2 weeks after completion of study treatment)
Population: All participants who received at least 1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks
Number analyzed (Participants) | 23 | 24 | 17 | 18 | 18
Percentage of Participants | 87.0 | 87.5 | 82.4 | 94.4 | 94.4

3. Primary Outcome: Percentage of Participants Discontinuing From Study Therapy Due to an AE
Description: as for outcome 2
Time Frame: Up to 16 weeks
Population: All participants who received at least 1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks
Number analyzed (Participants) | 23 | 24 | 17 | 18 | 18
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 5.6

4. Secondary Outcome: Percentage of Participants Achieving SVR24 (Sustained Virologic Response 24 Weeks After the End of All Study Therapy)
Description: The percentage of participants achieving SVR24 (i.e., HCV RNA < LLOQ 24 weeks after completing study treatment) was determined. Plasma HCV RNA levels were determined with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay, which has a LLOQ of 15 IU/mL.
Time Frame: Up to Week 40
Population: All randomized participants who received at least 1 dose of study drug, were not lost to follow-up for reasons unrelated to study treatment, and had SVR24 data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks
Number analyzed (Participants) | 23 | 21 | 16 | 17 | 16
Percentage of Participants | 91.3 [72.0 to 98.9] | 100.0 [83.9 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [80.5 to 100.0] | 93.8 [69.8 to 99.8]

ADVERSE EVENTS:
Time Frame: Up to 40 weeks
Description: All participants who received at least 1 dose of study drug are included.
Arm/Group | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 2/17 | 3/18 | 1/18
Other Adverse Events (participants affected / at risk) | 21/23 | 21/24 | 16/17 | 17/18 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks (N=23) | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks (N=24) | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks (N=17) | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks (N=18) | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks (N=18)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: HCV GT3 TN EBG/GZR+SOF+RBV 8 Weeks (N=23) | Arm 2: HCV GT3 TN EBG/GZR+SOF 12 Weeks (N=24) | Arm 3: HCV GT3 TE EBG/GZR+SOF 12 Weeks (N=17) | Arm 4: HCV GT3 TE EBG/GZR+SOF+RBV 12 Weeks (N=18) | Arm 5: HCV GT3 TE EBG/GZR+SOF 16 Weeks (N=18)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (3) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3) | 6 (7) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 6 (6) | 8 (10) | 6 (6) | 10 (10) | 6 (6)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3) | 3 (4) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 4 (5) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 7 (7) | 5 (7) | 11 (12) | 7 (7)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (2) | 3 (3) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.